CLINICAL TRIAL: NCT00027495
Title: Phase I Pharmacokinetic Trial of Curcuminoids Administered in a Capsule Formulation
Brief Title: Curcumin for the Prevention of Colon Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: CDR0000067916; P30CA046592 (NIH); CCUM-9941 (Other: University of Michigan Cancer Center PRC); NCI-P00-0144
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Cancer
Keywords: colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: curcumin

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. Curcumin may be effective in preventing the development of colon cancer.

PURPOSE: Phase I trial to determine the dose amount of curcumin that can be tolerated to help in preventing colon cancer in healthy men and women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of curcumin as a chemopreventive agent of colon cancer in healthy subjects.
* Determine if tolerable doses of this agent in uniformly milled formulation capsules are bioavailable in these subjects.
* Determine the pharmacokinetics of this agent and two metabolites at the MTD and next lower escalated dose in these subjects.

OUTLINE: This is a dose escalation study followed by a pharmacokinetic study.

Patients receive a single oral dose of curcumin followed by a standard fatty meal.

Cohorts of 3-6 patients receive escalating doses of curcumin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicities. Once the MTD is determined, additional patients are accrued to receive curcumin in the pharmacokinetic phase of the study.

Patients are followed at 24, 36, 48, and 72 hours.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for the dose escalation phase and then 12 additional patients will be accrued for the pharmacokinetic phase of this study within 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy men and women age 18 and over

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm3
* Hemoglobin greater than 12 g/dL
* Platelet count greater than 120,000/mm3

Hepatic:

* ALT/AST less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 1.5 times ULN
* Bilirubin less than 1.5 mg/dL

Renal:

* Creatinine less than 1.7 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior cancer except surgically resected basal cell or squamous cell skin cancer
* No history of peptic ulcer disease, gastrointestinal bleeding from gastric or duodenal ulcers, or gastrin secreting tumors
* No history of unreliability or noncompliance (missing pretreatment appointment more than twice)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 14 days since prior steroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 14 days since prior curcumin (turmeric) rich foods
* At least 14 days since prior nonsteroidal antiinflammatory drugs (NSAIDs)
* No chronic medications (i.e., daily for more than 28 days) except for oral contraceptives
* No concurrent coumadin or other anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12; Primary Completion 2004-02 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean E. Brenner, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States